CLINICAL TRIAL: NCT05994937
Title: Glycemic and Cardiometabolic Biomarker Improvements Associated With Reduction in Air Pollution Exposure
Brief Title: Cleaner Air for Lower Cardiometabolic Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-00755
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: PreDiabetes
Keywords: Air pollution; prediabetes; inflammation; cardiovascular disease prevention; blood sugar
MeSH Terms: conditions — Prediabetic State; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Portable Air Cleaner (PAC) Filtration (Experimental): High Efficiency Particulate Air (HEPA) filter will be left intact in the PAC for 4 weeks.
  Interventions: Device: PAC with HEPA filter intact
- Sham Portable Air Cleaner (PAC) Filtration (Sham Comparator): High Efficiency Particulate Air (HEPA) filter will be removed from the PAC for 4 weeks.
  Interventions: Device: PAC with HEPA filter removed

INTERVENTIONS:
Device: PAC with HEPA filter intact — A commercially available PAC with a true HEPA filter will be used. Unit will be placed in the bedroom and used continuously (24 hours/day) for a total of 4 weeks.
  Arms: Active Portable Air Cleaner (PAC) Filtration
Device: PAC with HEPA filter removed — Uses the same model as the experimental PAC that is identical in appearance and sound with the HEPA filter removed . Unit will be placed in the bedroom and used continuously (24 hours/day) for a total of 4 weeks.
  Arms: Sham Portable Air Cleaner (PAC) Filtration

SUMMARY:
The purpose of this interventional sham-controlled pilot study is to study the effects of using portable air cleaners (PACs) in outpatient adults with prediabetes. The primary aims are to determine the effect PAC's have on glycemic variability and the concentrations of circulating biomarkers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥18 years old
* Participant and members of household are reported to be non-smokers (defined as no household members are currently known to smoke cigarettes or use other tobacco products including e-cigarettes)
* Participant is to understand/speak English or Spanish
* Participant can understand study procedures and give informed consent
* Participant has prediabetes, defined as the absence of diabetes and any of the following: fasting plasma glucose 100-125 mg/dL, 2 hour plasma glucose of 140-199 mg/dL after 75 g oral glucose tolerance test, or A1c 5.7- 6.4%.
* Able to wear CGM for 2 two-week periods
* Able to participate in telephone or video conference for home equipment setup if needed
* Able to visit clinic for blood draws before and after the study period
* Do not intend to sleep anywhere outside of primary bedroom for more than 48 consecutive hours or a total of 7 days during the study period.
* Ability to lift, or access to assistance with lifting, 20 lb to set up air filter appliance in bedroom.
* Have not undergone major dietary change (such as change from usual diet to intermittent fasting or caloric restriction) in the past 2 weeks, and do not intend to during the study period

Exclusion Criteria:

* Participants who have diagnosed diabetes, or take antihyperglycemic medications
* Participants with known atherosclerotic disease: coronary artery disease, peripheral artery disease or history of cerebrovascular disease (stroke or Transient Ischemic Attack (TIA), carotid stenosis)
* Participants with known systemic inflammatory conditions (including but not limited to: inflammatory arthritis, vasculitides, inflammatory bowel diseases, cancer within past 5 years, Hashimoto's thyroiditis)
* Participants currently taking any anti-inflammatory medications or medications that target inflammatory cytokines
* Pregnancy: because blood glucose problems during pregnancy require intensive monitoring and lifestyle changes to protect the mother and fetus
* Participants with known or suspected Covid-19 in the prior 30 days
* Participants with post-covid sequelae (a.k.a "Long covid")
* Participants who are already utilizing HEPA filtration (PAC or within HVAC) in bedrooms

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Percent Change in A Continuous Glucose Monitor (CGM) Coefficient of Variation (CV) | Baseline, Week 4
  A CGM will be placed at baseline to continuously measure glucose, which will then be used to assess glycemic variability at the end of 4 weeks post-intervention. This outcome will be measured using the following equation: (([post-intervention]-[pre-intervention]))/([pre-intervention])*100%
Percent Change of C-reactive Protein (CRP) Biomarkers | Baseline, Week 4
  This outcome will be measured using the following equation: (([post-intervention]-[pre-intervention]))/([pre-intervention])*100%
Percent Change in Concentration of Interleukin-6 (IL-6) Biomarkers | Baseline, Week 4
  This outcome will be measured using the following equation: (([post-intervention]-[pre-intervention]))/([pre-intervention])*100%
Percent Change in Concentration of Tumor Necrosis Factor-alpha (TNFα) Biomarkers | Baseline, Week 4
  This outcome will be measured using the following equation: (([post-intervention]-[pre-intervention]))/([pre-intervention])*100%

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Newman, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Sharine.Wittkopp@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Sharine.Wittkopp@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.